CLINICAL TRIAL: NCT02115841
Title: Effect of Transcutaneous Nerve Stimulation on Primary Motor Cortex to Modulate Cortical Excitability and Hemodynamic Response During Implicit Motor Learning: A TMS and NIRS Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 102-2266A3
Record Dates: First submitted 2014-03-27; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Transcutaneous Nerve Stimulation
Keywords: Transcutaneous Nerve Stimulation; serial reaction time task; functional near infrared spectroscopy; transcranial magnetic stimulation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E1 (Experimental): Experiment 1 will measure the cortical excitability change after TENS intervention.
  Interventions: Device: "Enraf-Nonius" Muscle stimulator
- E2 (Experimental): Experiment 2 will measures implicit sequential motor task performance and cortical hemodynamic response using near infrared spectroscopy (NIRS) during motor execution. Cortical excitability will also be measured contemporary
  Interventions: Device: "Enraf-Nonius" Muscle stimulator

INTERVENTIONS:
Device: "Enraf-Nonius" Muscle stimulator — The order 15Hz TENS stimulation session and sham stimulation session will also be randomized.
  Other Names: Transcutaneous nerve stimulation

SUMMARY:
Noninvasive brain stimulation was recently gradually be emphasized. The electrical current applied on scalp can effective modulate cortical excitability. Forms of Stimulation included transcranial direct current stimulation(tDCS) and transcranial alternating stimulation(tACS). tDCS had been proved the effect of cortical excitability modulation. The polarization effect of direct current stimulation can modulation specific brain area and enhance motor performance. tACS was still controversial about the effect on cortical excitability. Previous study show that the frequency dependent excitatory or inhibitory effect on cortex. The possible mechanism was to affect brain oscillation status by provided different frequency of stimulation. Transcutaneous nerve stimulation (TENS) was common used on management of chronic pain. Peripheral nerve stimulation can enhance pain or sensory evoked potential was noted. Effect of low frequency TENS on central nervous is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Health Adult

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potential | Baseline,0 minute,30 minutes,60 minutes.
  Use single-pulse TMS to assess Motor evoked potential change.
Intracortical inhibition & Intracortical facilitation | Baseline,0 minute,30 minutes,60 minutes.
  Use paired-pulse TMS to record pre-test and post-test change.
Blood oxygen dependent level | Baseline,in experiment,0 minute,30 minutes,60 minutes.
  Use Near-infrared spectroscopy to record pre-test, in experiment, and post-test change
Implicit sequential motor task performance | Baseline,in experiment,0 minute,30 minutes,60 minutes.
  Change of Measure of Learning curve.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan